CLINICAL TRIAL: NCT03095079
Title: a Phase II Trial With Continuous Intravenous Infusion of Rh-endostatin in Combination With Dacarbazine and Cisplatin as the First Line Therapy for Metastatic Melanoma
Brief Title: Rh-endostatin in Combination With Dacarbazine and Cisplatin as the First Line Therapy for Metastatic Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of department of renal cancer and melanoma Affiliation: Beijing Cancer Hospital, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCH-MM-
Record Dates: First submitted 2017-03-20; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Melanoma
Keywords: endostar; dacarbazine; cisplatin
MeSH Terms: conditions — Melanoma | interventions — Endostatins; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EDP (Experimental): Dacarbazine,DTIC： 250 mg/m2/d，IV, d1-5 Cisplatin PDD：75 mg/m2，IV Endostar ENDO：15 mg/m2/d，CIV,d1~14
  Interventions: Drug: recombinant human endostatin

INTERVENTIONS:
Drug: recombinant human endostatin — Cisplatin:dose was based on patient's weight and could be adjusted for weight change,75 mg/m^2 by IV infusion separated in 3 different days Dacarbazine:250mg/m2,administered by intravenous (IV) infusion on the 1 to 5 day of each cycle
  Hr-endostatin:dose based on body surface area as 15mg/m2,continuous intravenous infusion from day 1 to day 14
  Other Names: endostar

SUMMARY:
The incidence of Melanoma is rapidly growthing,and in China,dacarbazine combined with cisplatin is conmendly used as the first-line chemotherapy of metastatic melanoma. But the response rate and survival results are very limited.This trial aim to add a safe and effective anti-angiogenesis drug,Human-recombinant endostatin,to find out a new strategy which may further extend the PFS and OS with a tolerated toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed melanoma with metastases and has no received any systemic treatment.
* 2.At least one measurable site (diameter≥1cm) of disease (RECIST 1.1).
* 3.Estimated life expectancy of 12 weeks or greater
* 4. ECOG performance status 0, 1
* 5.Adequate organ function
* 6.Without symptoms of brain metastases and stable in neuro-functions

Exclusion Criteria:

* 1. Pregnant or lactation women
* 2. Acute infections without control.
* 3. Heart disease history, cardiac function class≥NYHA II.
* 4. HIV positive or chronic HBV/HCV in active stage.
* 5. Brain metastases or primary tumor with positive symptoms
* 6. Need anti-epileptic treatments
* 7. Organ transplantation history
* 8. Hemorrhagic tendency or related history
* 9. Renal dialysis patients
* 10. Diagnosis of any second malignancy within the last 3 years, except for adequately treated.
* 11. Current treatment on another clinical trial
* 12. The other improper situations which investigator judged.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-12 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
progress-free survival(PFS) | From randomization up to 144 weeks
  Progression Free Survival is defined as the time from enrollment to the date of first documented disease progression or death from any cause

SECONDARY OUTCOMES:
Disease control rate(DCR) | From randomization up to 144 weeks
  CR+PR+SD
adverse events | From randomization up to 144 weeks
  Progression Free Survival is defined as the time from enrollment to the date of first documented disease progression or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Cui C, Mao L, Chi Z, Si L, Sheng X, Kong Y, Li S, Lian B, Gu K, Tao M, Song X, Lin T, Ren X, Qin S, Guo J. A phase II, randomized, double-blind, placebo-controlled multicenter trial of Endostar in patients with metastatic melanoma. Mol Ther. 2013 Jul;21(7):1456-63. doi: 10.1038/mt.2013.79. Epub 2013 May 14. PMID 23670576